CLINICAL TRIAL: NCT02268409
Title: An Open-Label Extension Study To Evaluate The Long-Term Effects Of ACE-536 In Patients With β-Thalassemia Previously Enrolled In Study A536-04
Brief Title: Extension Study to Evaluate the Safety and Efficacy of Luspatercept in Participants With β-Thalassemia Previously Enrolled in A536-04 (A536-06/MK-6143-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A536-06; A536-06 (Other: Acceleron); MK-6143-004 (Other: Merck); 2014-001281-94 (EudraCT Number)
Record Dates: First submitted 2014-10-06; First posted 2014-10-20 (Estimated); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-02

CONDITIONS: β-Thalassemia
MeSH Terms: interventions — luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Luspatercept Extension Population (Experimental): Participants receive luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants will receive the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
  Interventions: Drug: luspatercept

INTERVENTIONS:
Drug: luspatercept — subcutaneous injection
  Other Names: ACE-536; MK-6143

SUMMARY:
Study A536-06 (MK-6143-004) is an open-label extension study for participants previously enrolled in study A536-04 (NCT01749540), to evaluate the long-term safety and tolerability of luspatercept in adult participants with beta-thalassemia.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Completion of the treatment period in the base study A536-04.
* Females of child- bearing potential (defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy, or are not naturally postmenopausal ≥24 consecutive months) must have negative urine or blood pregnancy test prior to enrollment and use adequate birth control methods (abstinence, oral contraceptives, barrier method with spermicide, or surgical sterilization) during study participation and for 12 weeks following the last dose of study drug
* Males must agree to use a latex condom during any sexual contact with females of child-bearing potential during study participation and for 12 weeks following the last dose of study drug, even if he has undergone a successful vasectomy
* Participants must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of study drug
* Participants with treatment interruption (defined as participants who complete the end of study visit for study A536-04 and are ≥28 days post end of study visit) must also meet the following criteria:
* Mean hemoglobin concentration <10.0 g/dL of 2 measurements (not influenced by red blood cell [RBC] transfusion) (one performed within one day prior to first dose of study treatment and the other performed during the screening period [Day -28 to Day -1]) in non-transfusion dependent (NTD) participants
* Adequate folate levels or on folate therapy
* Platelet count ≥100 x 10^9/L and ≤1,000 x 10^9/L
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <3 x upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 x ULN
* Ejection fraction ≥50% by echocardiogram (ECHO) or multi-gated acquisition scan (MUGA)

Exclusion Criteria:

* Discontinuation/withdrawal from study A536-04 due to participant request, participant unwillingness or inability to comply with the protocol, pregnancy, use of prohibited medication (e.g., hydroxyurea), medical reason or adverse event, hypersensitivity reaction to the study drug, at the discretion of the sponsor, or loss to follow-up prior to completion of the treatment period
* Any clinically significant pulmonary (including pulmonary hypertension), cardiovascular, endocrine, neurologic, hepatic, gastrointestinal, infectious, immunological (including clinically significant allo- or auto-immunization) or genitourinary disease considered by the investigator as not adequately controlled prior to the first dose of study trearment
* Symptomatic splenomegaly
* Splenectomy within 56 days prior to the first dose of study treatment
* Major surgery (except splenectomy) within 28 days prior to the first dose of study treatment. Participants must have completely recovered from any previous surgery prior to the first dose of study treatment
* Participants receiving or planning to receive hydroxyurea treatment. Participants must not have had hydroxyurea within 90 days of the first dose of study treatment
* For participants with treatment interruption: Iron chelation therapy if initiated within 56 days prior to the first dose of study treatment
* Cytotoxic agents, systemic corticosteroids, immunosuppressants, or anticoagulant therapy such as warfarin or heparin within 28 days prior to the first dose of study treatment (prophylactic aspirin up to 100 mg/day and low molecular weight (LMW) heparin for superficial vein thrombosis (SVT) is permitted)
* Treatment with another investigational drug (including sotatercept [ACE-011]) or device, or approved therapy for investigational use ≤28 days prior to the first dose of study treatment, or if the half-life of the previous investigational product is known, within 5 times the half-life prior to the first dose of study treatment, whichever is longer at any time between the end of treatment of the base study A536-04 and the first dose of study treatment
* Known positive for human immunodeficiency virus (HIV), active infectious hepatitis B virus (HBV) or active infectious hepatitis C virus (HCV)
* Uncontrolled hypertension defined as systolic blood pressure (SBP) ≥150 mm mercury (Hg) or diastolic blood pressure (DBP) ≥100 mm Hg
* Known history of thromboembolic events ≥Grade 3 according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.0
* Pregnant or lactating females
* History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (7):
- Acceleron Investigative Site, Athens, Greece
- Italy (6):
  - Acceleron Investigative Site, Brindisi
  - Acceleron Investigative Site, Catania
  - Acceleron Investigative Site, Ferrara
  - Acceleron Investigative Site, Modena
  - Acceleron Investigative Site, Naples
  - Acceleron Investigative Site, Turin

REFERENCES:
- [Derived] Piga A, Longo F, Gamberini MR, Voskaridou E, Ricchi P, Caruso V, Pietrangelo A, Zhang X, Shetty JK, Attie KM, Tartaglione I. Long-term safety and erythroid response with luspatercept treatment in patients with beta-thalassemia. Ther Adv Hematol. 2022 Dec 5;13:20406207221134404. doi: 10.1177/20406207221134404. eCollection 2022. PMID 36505885
- [Derived] Piga A, Perrotta S, Gamberini MR, Voskaridou E, Melpignano A, Filosa A, Caruso V, Pietrangelo A, Longo F, Tartaglione I, Borgna-Pignatti C, Zhang X, Laadem A, Sherman ML, Attie KM. Luspatercept improves hemoglobin levels and blood transfusion requirements in a study of patients with beta-thalassemia. Blood. 2019 Mar 21;133(12):1279-1289. doi: 10.1182/blood-2018-10-879247. Epub 2019 Jan 7. PMID 30617198

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This extension study enrolled participants from the base study A536-04 (NCT01749540) following the last dose of luspatercept. Per protocol, participants were pooled from all doses received in the base study. Participants did not undergo an end of study visit in study A536-04 but instead were initiated immediately into the extension study.
Groups:
- Luspatercept Extension Population: Participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants received the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
Period: Overall Study
Arm/Group | Luspatercept Extension Population
Started | 51
Completed | 14
Not Completed | 37
Not completed — Reason for discontinuation not reported by the investigator | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 3
Not completed — Participation in study terminated by Sponsor | 25
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: All randomized participants who received ≥1 dose of study treatment
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Baseline Transfusion Status [Count of Participants; unit: Participants] — Participants were grouped for some endpoints in the extension study by transfusion dependence. Non-Transfusion dependence is defined as having received <4 units of red blood cells (RBCs) within 8 weeks prior to Cycle 1 Day 1. Transfusion dependence is defined as requiring ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to Cycle 1 Day 1).
  Participants
    Transfusion Dependent | 24
    Non-transfusion Dependent | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which did not necessarily have a causal relationship with the treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it was considered related to the study drug. The number of participants who experienced an AE is reported.
Time Frame: Up to approximately 68 months
Population: All participants that received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 51
Participants | 50

2. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due To an AE
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical investigation participant administered a study drug, which did not necessarily have a causal relationship with the treatment. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug whether or not it was considered related to the study drug. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to approximately 60 months
Population: All participants that received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 51
Participants | 5

3. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline Over a Rolling 8-week Interval
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL from baseline over an 8-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following RBC transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug. An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: All participants who received ≥1 dose of study treatment and received <4 units of RBCs within 8 weeks prior to the first dose of study drug and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- NTD Participants: NTD participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants received the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 77.8 [57.7 to 91.4]

4. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline Over a Rolling 12-week Interval
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL from baseline over a 12-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 77.8 [57.7 to 91.4]

5. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline During Weeks 13 to 24
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL from baseline measured during Weeks 13 to 24. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Weeks 13 to 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 59.3 [38.8 to 77.6]

6. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.0 g/dL From Baseline During Weeks 37 to 48
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.0 g/dL measured during Weeks 37 to 48. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of participants with a hemoglobin increase of ≥1.0 g/dL from baseline is presented.
Time Frame: Weeks 37 to 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 59.3 [38.8 to 77.6]

7. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline Over a Rolling 8-week Interval
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline over an 8-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline will is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 66.7 [46.0 to 83.5]

8. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline Over a Rolling 12-week Interval
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline over a 12-week interval compared to baseline. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 63.0 [42.4 to 80.6]

9. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline During Weeks 13 to 24
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline measured during Weeks 13 to 24. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline is presented.
Time Frame: Weeks 13 to 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 44.4 [25.5 to 64.7]

10. Secondary Outcome: Percentage of Non-transfusion Dependent (NTD) Participants With a Hemoglobin Increase of ≥1.5 g/dL From Baseline During Weeks 37 to 48
Description: An erythroid response in NTD participants was defined as a mean hemoglobin increase of ≥1.5 g/dL from baseline measured during Weeks 37 to 48. Baseline hemoglobin for NTD participants was the average of two or more measurements performed during the screening period of either the base study (A536-04) or the extension study (A536-06). Hemoglobin measurements within 2 weeks following red blood cell (RBC) transfusion were excluded from the analysis. NTD participants were participants who had received <4 units of RBCs within 8 weeks prior to the first dose of study drug. The percentage of participants with a hemoglobin increase of ≥1.5 g/dL from baseline is presented.
Time Frame: Weeks 37 to 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | NTD Participants
Number analyzed (Participants) | 27
Percentage of participants | 29.6 [13.8 to 50.2]

11. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥20% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 8-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a ≥20% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: All participants who received ≥1 dose of study treatment and received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug) and had data available for the analyses
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- TD Participants: TD participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants received the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 95.8 [78.9 to 99.9]

12. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥33% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 8-Week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a ≥33% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 95.8 [78.9 to 99.9]

13. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 8-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 95.8 [78.9 to 99.9]

14. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥20% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 12-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a ≥20% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 95.8 [78.9 to 99.9]

15. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥33% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 12-Week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a ≥33% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 83.3 [62.6 to 95.3]

16. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During a Rolling 12-week Interval
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 70.8 [48.9 to 87.4]

17. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥20% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 13 to 24
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a Weeks 13 to 24 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥20% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 13 to 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 58.3 [22.1 to 63.4]

18. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥33% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 13 to 24
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a Weeks 13 to 24 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥33% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 13 to 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 50.0 [29.1 to 70.9]

19. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 13 to 24
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during Weeks 13 to 24 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 13 to 24
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 33.3 [15.6 to 55.3]

20. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥20% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 37 to 48
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during Weeks 37 to 48 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥20% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 37 to 48
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 50.0 [29.1 to 70.9]

21. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥33% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 37 to 48
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during Weeks 37 to 48 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥33% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 37 to 48
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 50.0 [29.1 to 70.9]

22. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants With a ≥50% Reduction in Red Blood Cell (RBC) Transfusion Burden From Baseline During Weeks 37 to 48
Description: Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during Weeks 37 to 48 divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants with a ≥50% reduction in RBC transfusion burden from baseline is presented.
Time Frame: Weeks 37 to 48
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 33.3 [15.6 to 55.3]

23. Secondary Outcome: Percentage of Transfusion Dependent (TD) Participants Who Maintained Red Blood Cell (RBC) Transfusion Independence For ≥8 Weeks
Description: Transfusion independence for TD participants was defined as the percentage of participants who did not require RBC transfusion units (or milliliters) transfused for ≥8 weeks in the study after start of treatment. TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The percentage of participants who maintained transfusion independence for ≥8 weeks is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percentage of participants | 33.3 [15.6 to 55.3]

24. Secondary Outcome: Maximum Percent Change From Baseline in Red Blood Cell (RBC) Transfusions in Transfusion Dependent (TD) Participants Over 8 Weeks
Description: The reduction from baseline in red blood cell transfusions for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). An 8-week interval was defined as any consecutive 8 weeks during the study. The percentage change from baseline in RBC transfusions in TD participants is presented.
Time Frame: Any 8-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percent change | 80.4 (21.94)

25. Secondary Outcome: Maximum Percent Change From Baseline in Red Blood Cell (RBC) Transfusions in Transfusion Dependent (TD) Participants Over 12 Weeks
Description: The change from baseline in red blood cell transfusions for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). TD participants were participants who had received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug). A 12-week interval was defined as any consecutive 12 weeks during the study. The percentage change from baseline in RBC transfusions in TD participants is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TD Participants
Number analyzed (Participants) | 23
Percent change | 65.4 (25.62)

26. Secondary Outcome: Time To Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.0 g/dL Over a Rolling 12-week Interval
Description: Time to erythroid response was defined as the time from first dose to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.0 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The time to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.0 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: All participants who received ≥1 dose of study treatment and received <4 units of red blood cells (RBCs) within 8 weeks prior to the first dose of study drug and had data available for the analyses
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTD Participants
Number analyzed (Participants) | 21
Days | 13.6 (19.28)

27. Secondary Outcome: Time To Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.5 g/dL Over a Rolling 12-week Interval
Description: Time to erythroid response was defined as the time from first dose to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.5 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The time to the first date of any rolling 12-week window achieving a hemoglobin increase ≥1.5 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTD Participants
Number analyzed (Participants) | 17
Days | 104.0 (214.70)

28. Secondary Outcome: Time To Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥33% Over a Rolling 12-week Interval
Description: Time to erythroid response was defined as the time from first dose to the first date of any rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction compared to pretreatment of ≥33%. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The time to the first date of any rolling 12-week window achieving a red blood cell transfusion burden reduction compared to pretreatment of ≥33% is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: All participants who received ≥1 dose of study treatment and who have received ≥4 units of RBCs every 8 weeks (confirmed over 6 months prior to the first dose of study drug) and had data available for the analyses
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TD Participants
Number analyzed (Participants) | 20
Days | 14.6 (50.34)

29. Secondary Outcome: Time To Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥50% Over a Rolling 12-week Interval
Description: Time to erythroid response was defined as the time from first dose to the first date of any rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction compared to pretreatment of ≥50%. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The time to the first date of any rolling 12-week window achieving a red blood cell transfusion burden reduction compared to pretreatment of ≥50% is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TD Participants
Number analyzed (Participants) | 17
Days | 48.6 (107.53)

30. Secondary Outcome: Duration of Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.0 g/dL Over a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the starting date of the first rolling 12-week window achieving a hemoglobin increase of ≥1.0 g/dL to the last date of the last consecutive rolling 12-week window achieving a hemoglobin increase of ≥1.0 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The duration of response for participants achieving a hemoglobin increase ≥1.0 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTD Participants
Number analyzed (Participants) | 21
Days | 1147 (637.52)

31. Secondary Outcome: Duration of Erythroid Response for Non-transfusion Dependent (NTD) Participants Who Achieved a Hemoglobin Increase ≥1.5 g/dL Over a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the starting date of the first rolling 12-week window achieving a hemoglobin increase of ≥1.5 g/dL to the last date of the last consecutive rolling 12-week window achieving a hemoglobin increase of ≥1.5 g/dL. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The duration of response for participants achieving a hemoglobin increase ≥1.5 g/dL is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | NTD Participants
Number analyzed (Participants) | 17
Days | 969.3 (657.11)

32. Secondary Outcome: Duration of Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥33% Over a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the starting date of the first rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction compared to pretreatment of ≥33% to the last date of the last consecutive rolling 12-week window achieving a RBC transfusion burden reduction compared to pretreatment of ≥33%. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The duration of response for participants achieving a RBC transfusion burden reduction compared to pretreatment of ≥33% is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TD Participants
Number analyzed (Participants) | 20
Days | 487.5 (532.90)

33. Secondary Outcome: Duration of Erythroid Response for Transfusion Dependent (TD) Participants Who Achieved a Transfusion Burden Reduction of ≥50% Over a Rolling 12-week Interval
Description: Duration of erythroid response was defined as the time from the starting date of the first rolling 12-week window achieving a red blood cell (RBC) transfusion burden reduction compared to pretreatment of ≥50% to the last date of the last consecutive rolling 12-week window achieving a RBC transfusion burden reduction compared to pretreatment of ≥50%. When there were multiple disjointed intervals with response, the longest interval was used. Participants with response ongoing by the analysis cutoff day were censored. The duration of response for participants achieving a RBC transfusion burden reduction compared to pretreatment of ≥50% is presented.
Time Frame: Any 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | TD Participants
Number analyzed (Participants) | 17
Days | 462.5 (579.87)

34. Secondary Outcome: Mean Change From Baseline in Pre-transfusion Hemoglobin Levels in Transfusion Dependent (TD) Participants
Description: Pre-transfusion hemoglobin levels were calculated in TD participants. TD participants were participants who had received ≥4 units of red blood cells (RBC) every 8 weeks (confirmed over 6 months prior to the first dose of study drug). The baseline pre-transfusion hemoglobin level was an average of all hemoglobin values measured before the first dose of study drug given. The post-baseline pre-transfusion hemoglobin levels were calculated using the average of all hemoglobin values recorded before each transfusion that was required after the first dose of study drug was given. All hemoglobin levels measured within the 2 weeks following a red blood cell transfusion were excluded from the analysis. The change from baseline in pre-transfusion hemoglobin levels is presented.
Time Frame: Any 8 or 12-week interval during the study (up to approximately 68 months)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | TD Participants
Number analyzed (Participants) | 23
g/dL | -0.42 (0.59)

35. Secondary Outcome: Mean Change From Baseline in Hemoglobin Level Over Multiple Rolling 8-Week Intervals in Non-transfusion Dependent (NTD) Participants
Description: Mean change from baseline in hemoglobin levels was calculated for multiple rolling 8-week intervals in NTD participants. NTD participants were participants who had received <4 units of red blood cells (RBC) within 8 weeks prior to the first dose of study treatment. The baseline pre-transfusion hemoglobin level was an average of all hemoglobin values measured before the first dose of study drug given. The post-baseline hemoglobin level was taken after every rolling 8-week interval producing multiple values for the mean change from baseline in hemoglobin. The maximum change from baseline in hemoglobin level among the multiple rolling 8-week intervals is presented.
Time Frame: Baseline (prior to first dose of study drug) and multiple 8-week intervals during the study (up to approximately 68 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NTD Participants
Number analyzed (Participants) | 26
g/dL | 1.9 (1.04)

36. Secondary Outcome: Mean Change From Baseline in Hemoglobin Level Over Multiple Rolling 12-Week Intervals in Non-transfusion Dependent (NTD) Participants
Description: Mean change from baseline in hemoglobin levels was calculated for multiple rolling 12-week intervals in NTD participants. NTD participants were participants who had received <4 units of red blood cells (RBC) within 8 weeks prior to the first dose of study treatment. The baseline pre-transfusion hemoglobin level was an average of all hemoglobin values measured before the first dose of study drug given. The post-baseline hemoglobin level was taken after every rolling 12-week interval producing multiple values for the mean change from baseline in hemoglobin. The maximum change from baseline in hemoglobin level among the multiple rolling 12-week intervals is presented.
Time Frame: Baseline (prior to first dose of study drug) and multiple 12-week intervals during the study (up to approximately 68 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | NTD Participants
Number analyzed (Participants) | 26
g/dL | 1.8 (1.06)

37. Secondary Outcome: Percent Change From Baseline in Transfusion Burden Over Multiple Rolling 8-Week Intervals in Transfusion Dependent (TD) Participants
Description: Percent change from baseline in transfusion burden was calculated for multiple rolling 8-week intervals in TD participants. TD participants were participants who had received ≥4 units of red blood cells (RBC) every 8 weeks (confirmed over 6 months prior to the first dose of study drug). Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during an 8-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 8 weeks prior to the start of treatment (baseline). The post-baseline transfusion burden was calculated after every rolling 8-week interval producing multiple values for the percent change from baseline in transfusion burden. The maximum percent change from baseline in transfusion burden among the multiple rolling 8-week intervals is presented.
Time Frame: as for outcome 35
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TD Participants
Number analyzed (Participants) | 24
Percent change | 80.4 (21.94)

38. Secondary Outcome: Percent Change From Baseline in Transfusion Burden Over Multiple Rolling 12-Week Intervals in Transfusion Dependent (TD) Participants
Description: Percent change from baseline in transfusion burden was calculated for multiple rolling 12-week intervals in TD participants. TD participants were participants who had received ≥4 units of red blood cells (RBC) every 8 weeks (confirmed over 6 months prior to the first dose of study drug). Transfusion burden for TD participants was defined as the ratio of RBC transfusion units (or milliliters) transfused during a 12-week interval divided by the duration of that interval compared to the ratio of RBC transfusion units 12 weeks prior to the start of treatment (baseline). The post-baseline transfusion burden was calculated after every rolling 12-week interval producing multiple values for the percent change from baseline in transfusion burden. The maximum percent change from baseline in transfusion burden among the multiple rolling 12-week intervals is presented.
Time Frame: as for outcome 36
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | TD Participants
Number analyzed (Participants) | 23
Percent change | 65.4 (25.62)

39. Secondary Outcome: Percent Change From Baseline to End of Treatment in Erythropoietin
Description: Blood samples were collected at pre-specified time intervals to determine erythropoietin. The percent change from baseline in mean concentration of erythropoietin was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for erythropoietin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Non-transfusion Dependent (NTD) Participants: NTD participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants received the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
- Transfusion Dependent (TD) Participants: TD participants received luspatercept 0.6, 0.8, 1.0, or 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years). Participants received the highest tolerated dose level of luspatercept that they were assigned in the base study unless a dose modification was required.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 22 | 20
Percent change | 10.18 (66.02) | 105.15 (179.22)

40. Secondary Outcome: Percent Change From Baseline to End of Treatment in Reticulocyte Count
Description: Blood samples were collected at pre-specified time intervals to determine reticulocyte count. The percent change from baseline in reticulocyte count was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for reticulocyte analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 20 | 18
Percent change | 32.46 (47.62) | 220.90 (539.20)

41. Secondary Outcome: Percent Change From Baseline to End of Treatment in Nucleated Red Blood Cell (nRBC) Count
Description: Blood samples were collected at pre-specified time intervals to determine nRBC count. The percent change from baseline in nRBC count was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for nRBC analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 13 | 12
Percent change | 52.15 (96.24) | 579.58 (867.44)

42. Secondary Outcome: Percent Change From Baseline to End of Treatment in Soluble Transferrin Receptor
Description: Blood samples were collected at pre-specified time intervals to determine soluble transferrin receptor. The percent change from baseline in mean concentration of soluble transferrin receptor was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for soluble transferrin receptor analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 22 | 20
Percent change | 3.3 (23.42) | 53 (56.29)

43. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Ferritin
Description: Blood samples were collected at pre-specified time intervals to determine serum ferritin. The percent change from baseline in mean concentration of serum ferritin was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for serum ferritin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 22 | 20
Percent change | -22.8 (38.65) | -22.4 (52.95)

44. Secondary Outcome: Percent Change From Baseline to End of Treatment in Percent Transferrin (Iron) Saturation
Description: Blood samples were collected at pre-specified time intervals to determine percent transferrin (iron) saturation. The percent change from baseline in mean concentration of percent transferrin (iron) saturation was measured. Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for percent transferrin (iron) saturation analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 22 | 20
Percent change | 10.1 (44.63) | -2.6 (43.95)

45. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Transferrin
Description: Blood samples were to be collected at pre-specified time intervals to determine serum transferrin. Baseline was pre-specified to be the last measurement prior to the first dose of study drug. Per protocol, the analysis was planned to be presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: No data were collected for Percent Change From Baseline to End of Treatment in Serum Transferrin.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 0 | 0

46. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Iron
Description: Blood samples were to be collected at pre-specified time intervals to determine serum iron. Baseline was pre-specified to be the last measurement prior to the first dose of study drug. Per protocol, the analysis was planned to be presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: No data were collected for Percent Change From Baseline to End of Treatment in Serum Iron.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Hepcidin
Description: Blood samples were to be collected at pre-specified time intervals to determine serum hepcidin. Baseline was pre-specified to be the last measurement prior to the first dose of study drug. Per protocol, the analysis was planned to be presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: No data were collected for Percent Change From Baseline to End of Treatment in Serum Hepcidin.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 0 | 0

48. Secondary Outcome: Percent Change From Baseline to End of Treatment in Serum Total Iron Binding Capacity (TIBC)
Description: Blood samples were to be collected at pre-specified time intervals to determine serum total iron binding capacity. Baseline was pre-specified to be the last measurement prior to the first dose of study drug. Per protocol, the analysis was planned to be presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: No data were collected for Percent Change From Baseline to End of Treatment in Serum TIBC.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 0 | 0

49. Secondary Outcome: Percent Change From Baseline to End of Treatment in Non-transferrin Bound Iron (NTBI)
Description: Blood samples were to be collected at pre-specified time intervals to determine serum non-transferrin bound iron. Baseline was pre-specified to be the last measurement prior to the first dose of study drug. Per protocol, the analysis was planned to be presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: No data were collected for Percent Change From Baseline to End of Treatment in NTBI.
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 0 | 0

50. Secondary Outcome: Percent Change From Baseline to End of Treatment in Total Bilirubin
Description: Blood samples were collected at pre-specified time intervals to determine total bilirubin. The percent change from baseline in total bilirubin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for total bilirubin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 39
Percent change | 13.3 (31.69)

51. Secondary Outcome: Percent Change From Baseline to End of Treatment in Indirect Bilirubin
Description: Blood samples were collected at pre-specified time intervals to determine indirect bilirubin. The percent change from baseline in indirect bilirubin was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for indirect bilirubin analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 39
Percent change | 46.1 (169.03)

52. Secondary Outcome: Percent Change From Baseline to End of Treatment in Lactate Dehydrogenase (LDH)
Description: Blood samples were collected at pre-specified time intervals to determine LDH. The percent change from baseline in LDH was measured. Baseline was the last measurement prior to the first dose of study drug.
Time Frame: Baseline (prior to first dose of study drug) and End of Treatment (up to Day 1807)
Population: All participants who received ≥1 dose of study treatment and had data available for LDH analyses
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 41
Percent change | 13.6 (57.8)

53. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC <3 mg/g Dry Weight Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC <3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC <3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 3 | 7
mg/g dry weight | 0.02 (0.055) | 0.72 (0.864)

54. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC ≥3 mg/g Dry Weight Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC ≥3 mg/g dry weight was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC ≥3 mg/g dry weight, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 10 | 6
mg/g dry weight | -1.64 (2.068) | -3.41 (3.434)

55. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC <3 mg/g Dry Weight, Who Have Used Iron Chelation Therapy (ICT), Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC <3 mg/g dry weight and who have used ICT within 84 days prior to the first dose of study drug or during the study treatment period was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC <3 mg/g dry weight, who have used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 1 | 7
mg/g dry weight | -0.03 (NA) — Standard deviation cannot be calculated on data from 1 participant. | 0.72 (0.864)

56. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC ≥3 mg/g Dry Weight, Who Have Used Iron Chelation Therapy (ICT), Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC ≥3 mg/g dry weight and who have used ICT within 84 days prior to the first dose of study drug or during the study treatment period was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC ≥3 mg/g dry weight, who have used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 7 | 5
mg/g dry weight | -1.97 (2.287) | -4.38 (2.788)

57. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC <3 mg/g Dry Weight, Who Have Not Used Iron Chelation Therapy (ICT), Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC <3 mg/g dry weight and who have not used ICT within 84 days prior to the first dose of study drug or during the study treatment period was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC <3 mg/g dry weight, who have not used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 2 | 0
mg/g dry weight | 0.04 (0.056) |

58. Secondary Outcome: Change From Baseline in Liver Iron Concentration (LIC) For Participants With Baseline LIC ≥3 mg/g Dry Weight, Who Have Not Used Iron Chelation Therapy (ICT), Measured After 18 Months and Up to 60 Months of Treatment
Description: Blood samples were collected at pre-specified time intervals to determine LIC. The change from baseline in mean LIC for participants with baseline LIC ≥3 mg/g dry weight and who have not used ICT within 84 days prior to the first dose of study drug or during the study treatment period was measured using magnetic resonance imaging (MRI). Baseline was the last measurement prior to the first dose of study drug. Per protocol, the analysis was presented by transfusion status (non-transfusion and transfusion dependent).
Time Frame: Baseline (prior to first dose of study drug) and up to approximately 60 Months
Population: All participants with baseline LIC ≥3 mg/g dry weight, who have not used ICT, who received ≥1 dose of study treatment, and had data available for the analyses
Measure: Mean (Standard Deviation); unit: mg/g dry weight
Arm/Group | Non-transfusion Dependent (NTD) Participants | Transfusion Dependent (TD) Participants
Number analyzed (Participants) | 3 | 1
mg/g dry weight | -0.88 (1.514) | 1.4 (NA) — Standard deviation cannot be calculated on data from 1 participant.

59. Secondary Outcome: Serum Concentration of Luspatercept
Description: Blood samples were collected at multiple time points to determine the serum concentration of luspatercept. Serum concentrations that were below the limit of quantitation (LOQ) of the assay prior to the first dose were assigned a numerical value of zero. Post-treatment serum concentrations that were below the LOQ of the assay were treated as missing. Serum concentrations assigned a value of missing were omitted from the analysis. The LOQ of the assay was 50 ng/mL.
Time Frame: Predose and Postdose Days 1, 8, 22, 169, 176, 190, 337, and 344
Population: All participants who received ≥1 dose of study treatment and had data available for serum concentration analyses
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Luspatercept Extension Population
Number analyzed (Participants) | 51
ng/mL
  Day 1: number analyzed (Participants) | 26
  Day 1 | 72.23 (303.23)
  Day 8 | 6096 (2853.45)
  Day 22 | 2756.78 (1635.41)
  Day 169: number analyzed (Participants) | 39
  Day 169 | 3929.49 (1614.99)
  Day 176: number analyzed (Participants) | 39
  Day 176 | 8675.97 (3039.6)
  Day 190: number analyzed (Participants) | 40
  Day 190 | 4008.2 (2004.9)
  Day 337: number analyzed (Participants) | 34
  Day 337 | 3985.94 (2018.04)
  Day 344: number analyzed (Participants) | 31
  Day 344 | 8768.84 (3334.63)

ADVERSE EVENTS:
Time Frame: Up to approximately 68 months
Description: All-cause mortality was reported on all randomized participants. Serious and non-serious adverse events (AEs) were reported on all participants who received ≥1 dose of study treatment. Data are presented by the dose of luspatercept that was administered at the time when the AE or death occurred.
Groups:
- Luspatercept 0.6 mg/kg: Participants received luspatercept 0.6 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 0.8 mg/kg: Participants received luspatercept 0.8 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 1.0 mg/kg: Participants received luspatercept 1.0 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
- Luspatercept 1.25 mg/kg: Participants received luspatercept 1.25 mg/kg administered by subcutaneous injection on Day 1 of each 21-day cycle for up to 87 cycles (up to approximately 5 years).
Arm/Group | Luspatercept 0.6 mg/kg | Luspatercept 0.8 mg/kg | Luspatercept 1.0 mg/kg | Luspatercept 1.25 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/49 | 0/41 | 1/38
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/49 | 2/41 | 3/38
Other Adverse Events (participants affected / at risk) | 2/2 | 39/49 | 30/41 | 37/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.6 mg/kg (N=2) | Luspatercept 0.8 mg/kg (N=49) | Luspatercept 1.0 mg/kg (N=41) | Luspatercept 1.25 mg/kg (N=38)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Luspatercept 0.6 mg/kg (N=2) | Luspatercept 0.8 mg/kg (N=49) | Luspatercept 1.0 mg/kg (N=41) | Luspatercept 1.25 mg/kg (N=38)
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (11)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (7)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (4)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2) | 7 (9)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 9 (20)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 8 (8) | 4 (7) | 14 (30)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 5 (26)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (7) | 5 (6) | 6 (13)
Toothache (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (8) | 2 (2) | 8 (10)
Asthenia (General disorders) | 0 (0) | 13 (24) | 6 (10) | 18 (61)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Influenza like illness (General disorders) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
Injection site pain (General disorders) | 0 (0) | 2 (2) | 2 (3) | 4 (4)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 0 (0) | 4 (7)
Pyrexia (General disorders) | 1 (1) | 18 (27) | 10 (20) | 21 (59)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 7 (11)
Influenza (Infections and infestations) | 0 (0) | 5 (6) | 4 (4) | 11 (21)
Nasopharyngitis (Infections and infestations) | 0 (0) | 5 (6) | 1 (1) | 7 (11)
Oral herpes (Infections and infestations) | 0 (0) | 2 (4) | 0 (0) | 4 (9)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 2 (2) | 7 (23)
Rhinitis (Infections and infestations) | 0 (0) | 4 (5) | 1 (1) | 12 (24)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 6 (11)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 2 (3)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (6) | 0 (0) | 3 (6)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 10 (15) | 4 (9) | 15 (31)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (16) | 3 (3) | 12 (29)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 18 (30) | 8 (14) | 16 (48)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (28) | 4 (6) | 9 (35)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (11) | 3 (4) | 16 (26)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (5)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 10 (24)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 3 (7) | 4 (6) | 9 (23)
Headache (Nervous system disorders) | 2 (9) | 14 (72) | 9 (10) | 19 (122)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Priapism (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (8) | 2 (2) | 12 (38)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 7 (32)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (10) | 6 (9) | 14 (43)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 6 (10)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (7)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (25)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (8) | 0 (0) | 2 (5)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Systolic hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication or disclosure of study results will be permitted except as specified in a separate, written, agreement between the sponsor and the investigator(s).

DOCUMENTS (2):
  • Study Protocol (2019-03-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT02268409/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT02268409/SAP_001.pdf